CLINICAL TRIAL: NCT02346084
Title: CHARM-03: A Randomized, Open Label, Crossover Phase 1 Safety and Pharmacokinetic Study of Oral Maraviroc and Maraviroc 1% Gel Administered Rectally and Vaginally to HIV-1 Seronegative Adults
Brief Title: Safety and Pharmacokinetic Study of Oral Maraviroc and Maraviroc 1% Gel in HIV-1 Seronegative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Maraviroc 1% Gel (Charm); AI082637 (Other: DAIDS)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; Tablets; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Female Participants - Arms 1A through 9A (Experimental): Female Participants 9 Arms (1A through 9A) 3 Product Sequences
  Product Sequence 1 Rx1- MVC tablet PO Rx2- MVC 1% gel PR Rx3- MVC 1% gel PV
  Product Sequence 2 Rx1- MVC 1% gel PR Rx2- MVC 1% gel PV Rx3- MVC tablet PO
  Product Sequence 3 Rx1- MVC 1% gel PV Rx2- MVC tablet PO Rx3- MVC 1% gel PR
  3 Biopsy Schedules D8- (~2-hr after the 8th dose) D9- (~24-hr after the 8th dose) D10- (~48-hr after the 8th dose)
  Interventions: Drug: Maraviroc 300 mg tablet (PO) and Maraviroc 1% gel (PR and PV)
- Male Participants - Arms 1B through 4B (Experimental): Male Participants 4 Arms (1B through 4B) 2 Product Sequences 2 biopsy schedules
  Product Sequence 1 Rx1- MVC tablet PO Rx2- MVC 1% gel PR
  Product Sequence 2 Rx1- MVC 1% gel PR Rx2- MVC tablet PO
  Biopsy Schedule D8- (~2-hr after the 8th dose) D10- (~48-hr after the 8th dose)
  Interventions: Drug: Maraviroc 300 mg tablet (PO) and Maraviroc 1% gel (PR and PV)

INTERVENTIONS:
Drug: Maraviroc 300 mg tablet (PO) and Maraviroc 1% gel (PR and PV) — Tablets: daily 300 mg oral maraviroc, Selzentry®,(MVC) for 8 consecutive days Gel: daily rectally administered 1% MVC gel for 8 daily consecutive days Female Participants - will receive an additional third regimen of daily vaginally administered MVC 1% gel for 8 consecutive days.
  Each treatment regimen will be followed by a washout period of 14 to 21 days.
  Participants will also be randomized to a biopsy sampling schedule (i.e., D8, D9, or D10 sampling).
  Other Names: Tablet - Selzentry®, (MVC)

SUMMARY:
The purpose of the study is to evaluate the safety, acceptability, and PK/PD profile of maraviroc gel following rectal and vaginal administration. The study also includes oral exposure to maraviroc.

DETAILED DESCRIPTION:
Trail 11991 is a Phase 1 randomized, open label, single-site trial. Approximately 19 participants (9 female, 10 male) will be randomized to the 9 female study arms and 4 male study arms with 1-3 participants per arm. The randomization will be completed for the product sequence and the timing of tissue sample collection.

All participants will receive both study products by multiple routes of administration (i.e., PO, PR, [and PV for female participants]), and they will be randomized to the order of product sequence and specimen sampling schedule. The male participants will receive oral and rectal MVC and the female participants will receive oral, rectal, and vaginal MVC, in randomized sequence.

Participant accrual will take approximately 6 months. Male participants will be on study for approximately 9 to 12 weeks. Female participants will be on study for approximately 12 to 16 weeks. The total duration of the study will be approximately 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 through 45 at screening, verified per site SOP
2. Male participants, born male; female participants, born female.
3. Willing and able to communicate in English
4. Willing and able to provide written informed consent to take part in the study
5. Willing and able to provide adequate locator information, as defined in site SOP
6. Availability to return for all study visits, barring unforeseen circumstances
7. Understands and agrees to local sexually transmitted infection (STI) reporting requirements
8. HIV-1 seronegative at screening and enrollment
9. Must be in general good health in the opinion of the investigator
10. Willing to abstain from insertion of anything in the rectum (e.g., penis, sex toy, medication, enemas) 72 hours before all rectal sampling visits and 72 after rectal biopsy visits
11. Must agree to use study-provided condoms for insertive and receptive intercourse, whether vaginal or anal, for the duration of the study
12. Must agree not to participate in other concurrent interventional and/or drug trials

    Female participants must meet the following criteria:
13. Per participant report at Screening:

    1. Not pregnant or breastfeeding
    2. Regular menstrual cycles with at least 21 days between menses
    3. Satisfactory cervical Pap result in the 24 calendar months prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines in the 12 calendar months prior to Enrollment.
    4. Willing to abstain from vaginal insertion of anything (e.g., penis, sex toy, tampon, medication, douche) for 72 hours before all cervicovaginal sampling visits and 1 week after cervical biopsy visits
14. Per participant report at Enrollment:

    e) Using an effective method of contraception and intending to continue use of an effective method for the duration of study participation. Effective methods include hormonal methods (except contraceptive vaginal rings), intrauterine device (IUD) inserted at least 28 days prior

    Male participants must meet the following criteria:
15. Per participant report at Enrollment:

    1. Using an effective method of contraception and intending to continue use of an effective method for the duration of study participation. Effective methods include male condoms, surgical sterilization, being a man who identifies as a man who has sex with men exclusively, sexually abstinent for the past 90 days, and/or female partner use of hormonal contraception, intrauterine device [IUD], or surgical sterilization

Exclusion Criteria:

1. Undergoing or completed gender reassignment
2. Participant reports any of the following at Screening:

   1. Post-exposure prophylaxis for HIV exposure within 4 weeks prior to screening
   2. Reports history of unprotected insertive or receptive anal intercourse within 3 months prior to screening
   3. History of sexually transmitted disease in the last 3 months
   4. Known HIV-infected partners
   5. Non-therapeutic injection drug use in the 12 months prior to screening
   6. History of recurrent urticaria
   7. Allergy to soy, soybeans, peanuts, methylparaben, propylparaben, or sorbic acid
   8. Use of antiretroviral medications with activity against HIV within the 4 weeks prior to the Enrollment
   9. Use of systemic immunomodulatory medications within the 4 weeks prior to the Enrollment
   10. Use of vaginally or rectally administered medications or products (including condoms) containing Nonoxynol-9 (N-9) within the 4 weeks prior to the Enrollment
   11. Participating in another research study involving drugs or medical devices within the 4 weeks prior to the Enrollment
   12. Has plans to relocate away from the study site area during the period of study participation
3. Per participant report at screening, anticipated use and/or unwillingness to abstain from the following medications during the period of study participation:

   1. Heparin, including Lovenox® (enoxaparin sodium)
   2. Warfarin
   3. Plavix® (clopidogrel bisulfate)
   4. Any other drugs that are associated with increased likelihood of bleeding following mucosal biopsy (e.g., daily high dose aspirin (> than 81 mg), NSAIDs, or Pradaxa®)
   5. Rectally or vaginally administered medications (including over-the-counter products)
   6. Use of potent CYP3A inhibitors (e.g., ketoconazole and clarithromycin), and CYP3A inducers (e.g., anti-convulsants and St.John's wort)
   7. Multiple dose dexamethasone
   8. Antiretroviral medications with activity against HIV
4. History of significant gastrointestinal bleeding in the opinion of the investigator
5. Abnormalities of the cervical, vaginal, or colorectal mucosa, or significant symptom(s), which in the opinion of the clinician represents a contraindication to protocol-required biopsies (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids).
6. Body mass index (BMI) < 18 or > 35 kg/m2
7. At screening: participant-reported symptoms, and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current CDC guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include symptomatic bacterial vaginosis, symptomatic vaginal candidiasis, other vaginitis, trichomoniasis, Chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, pelvic inflammatory disease, genital sores or ulcers, cervicitis, or symptomatic genital warts requiring treatment. Note that an HSV-1 or HSV-2 seropositive diagnosis with no active lesions is allowed, since treatment is not required. Note: In cases of genital GC/CT identified at screening, one re-screening 2 months after screening visit will be allowed
8. Has any of the following laboratory abnormalities at Screening:

   CHARM-03, Version 1.0 28 31st July 2014
   1. Hemoglobin < 10.0 g/dL
   2. Platelet count less than 100,000/mm3
   3. White blood cell count < 2,000 cells/mm3 or > 15,000 cells/mm3
   4. Calculated creatinine clearance ≤ 70 mL/minute using the Cockcroft-Gault equation
   5. Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 2.5× the site laboratory ULN
   6. Total bilirubin > 2.5 ULN
   7. ≥ +1 glucose or +2 protein on urinalysis (UA)
   8. International Normalized Ratio (INR) test > 1.5× the site laboratory upper limit of normal (ULN)
   9. Positive for Hepatitis B surface antigen (HBsAg)
   10. Positive for Hepatitis C antibody (HCV Ab)
   11. CCR5 Δ 32 homozygous or heterozygous
9. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease In addition to the criteria listed above, female participants will be excluded if they meet any of the following criteria:
10. Participant reports any of the following at Screening:

    1. Last pregnancy outcome or gynecological surgery 90 days or less prior to screening
    2. Intends to become pregnant during the period of study participation
    3. Chronic and/or recurrent symptomatic vaginal candidiasis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
AEs Grade 2 or higher as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events | Female participants will be on study for approximately 12 to 16 weeks. Male participants will be on study for approximately 9 to 12 weeks. The total duration of the study will be approximately 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ian McGowan, MD, PhD, FRCP, Study Chair — Magee-Women's Research Institute
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] McGowan IM, Chawki S, Hendrix CW, Anton PA, Marzinke MA, Brand RM, Engstrom JC, Rohan LC, Abebe KZ, Richardson-Harman N, Siegel A, Reinhart A, Steytler J, Stall R, Spiegel H, Chen B, Achilles SL, Jacobson CE, Khanukova E, Cranston RD. A Randomized, Open-Label, Crossover Phase 1 Safety and Pharmacokinetic Study of Oral Maraviroc and Maraviroc 1% Gel (the CHARM-03 Study). AIDS Res Hum Retroviruses. 2022 Apr;38(4):269-278. doi: 10.1089/AID.2021.0096. Epub 2021 Sep 14. PMID 34384282